CLINICAL TRIAL: NCT01513161
Title: A 14 Day, Multi-center, Randomized, Double Blinded, Placebo-controlled, Parallel Group, Fixed Dose, Phase III Clinical Trial to Assess the Efficacy and Safety of TRK-820 in Treating Conventional-treatment-resistant Pruritus in Patients Receiving Hemodialysis
Brief Title: Efficacy and Safety Study of TRK-820 to Treat Conventional-treatment-resistant Pruritus in Patients Receiving Hemodialysis
Acronym: TRK-820
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Collaborators: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TRK-820_PRU_III_2007
Record Dates: First submitted 2010-11-23; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Conventional-treatment-resistant Pruritus in Patients Receiving Hemodialysis
Keywords: pruritus
MeSH Terms: conditions — Pruritus | interventions — TRK 820

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TRK-820 5μg (Active Comparator): Taking TRK-820 5μg(two 2.5μg capsules) by oral route once daily for 14 days
  Interventions: Drug: nalfurafine hydrochloride (TRK-820)
- TRK-820 2.5μg (Active Comparator): Taking TRK-820 2.5μg(one 2.5μg capsule & one placebo capsule)by oral route once daily for 14 days
  Interventions: Drug: nalfurafine hydrochloride (TRK-820)
- Placebo (Placebo Comparator): Taking Placebo(two placebo capsule) by oral route once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nalfurafine hydrochloride (TRK-820) — Soft capsule containing 2.5ug nalfurafine hydrochloride. Start with 2.5ug of oral administraion once daily, and can be increased up to 5ug if necessary.
  Arms: TRK-820 2.5μg; TRK-820 5μg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether nalfurafine hydrochloride is effective and safe in the treatment for conventional-treatment-resistant pruritus in patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

[At the time of obtaining the consent form]

* Chronic renal failure patients who regularly receive hemodialysis three times a week and are not likely to have a serious treatment change or acute symptoms during the study period
* Patients who received both of the drug pruritus treatments in section 1 and 2 below within one year before the day of singing consent form

  1. Systemic therapy of more than two consecutive weeks depending on antihistamine or antiallergic drugs falling under "prescription drugs with indication of pruritus" (oral drugs, injections, etc.)
  2. Local therapy depending on "prescription drugs with indication of pruritus" (ointment, etc.) or a moisturizer prescribed by a doctor (topical preparation, etc.)
* Patients for whom all the conventional pruritus treatments in section (2) are not enough
* Patients aged 20 years or older at time of signing the consent form

[At the time of enrollment]

* Patients whose VAS scores are measured both after breakfast and dinner for five days or more of the last 7 days of the predose observation period and whose mean of whichever the higher VAS scores after breakfast or dinner is ≥50 mm
* Patients whose whichever the higher VAS score after breakfast or dinner for the last 7 days during the preliminary observation day (measured VAS score if one is missing) is more than ≥20 mm for five days or more
* Patients who are judged to have pruritus both during the day and at night for more than two days based on the Shiratori's severity criteria assessed by the subject at days of fifth and sixth hemodialysis and the day of hemodialysis after the completion of the predose observation period, and whose whichever the higher pruritis score measured during the day or at night is 3 (moderate) for two days or more

Exclusion Criteria:

* Patients with malignant tumor
* Patients with depression, schizophrenia or dementia as complications
* Patients who currently have Child-pugh class B or C hepatic cirrhosis as complications
* Patients with clinically significant hepatic or cardiovascular diseases which cannot be controlled by diet or drug therapy
* Patients who currently have the following heart diseases: life-threatening arrhythmia; unstable angina or myocardiac infarction within 6 months; PCI or CABG within 6 months; NYHA class III or IV congestive heart failure
* Patients with atopic dermatitis or chronic urticaria as complications
* Patients who are allergic to opioid drugs
* Patients with dependence on drug or alcohol
* Patients who received phototherapy for pruritus within one month before signing the consent form
* Patients who participated in the study of TRK-820 and received the study drug or who were already enrolled in this study
* Patients who participated in other clinical studies (including the ones using artificial kidney and medical equipment), and received the study drug or treatment with clinical equipment within one month before signing the consent form
* Pregnant women, lactating women and patients of childbearing potential who do not use contraceptive methods
* Patients who cannot report VAS scores by their own for any reason at the principal investigator or study personnel's discretion
* Patients whose complications or history can impact the results of this study at the principal investigator or subinvestisator's discretion
* Other patients who are not proper to participate in this study at the principal investigator or study personnel's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in pruritus degree measured by VAS(Visual Analogue Scale) score | 4 weeks (2 weeks measurement with only conventional treatment + 2 weeks measurement with conventional treatment & investigational products)

SECONDARY OUTCOMES:
Changes in Shiratori's severity scores assessed by the subject. | 4 weeks (2 weeks measurement with only conventional treatment + 2 weeks measurement with conventional treatment & investigational products)

CONTACTS AND LOCATIONS:
Overall Officials: Suhng Gwon Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SKchemicals Investigational Site, Seoul, South Korea

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264